CLINICAL TRIAL: NCT01228591
Title: Pilot Dispensing Evaluation of a Plus Power Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR-1636BB
Record Dates: First submitted 2010-10-22; First posted 2010-10-26 (Estimated); Results first posted 2014-02-03 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2015-05

CONDITIONS: Hyperopia
MeSH Terms: conditions — Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acuvue Advance Plus/ Acuvue Advance (Other): Acuvue Advance Plus contact lenses worn first period and Acuvue Advance contact lenses worn second.
  Interventions: Device: Acuvue Advance Plus; Device: Acuvue Advance
- Acuvue Advance/Acuvue Advance Plus (Other): Acuvue Advance contact lenses worn first period and Acuvue Advance Plus contact lenses worn second.
  Interventions: Device: Acuvue Advance Plus; Device: Acuvue Advance

INTERVENTIONS:
Device: Acuvue Advance Plus — Silicone hydrogel contact lens.
Device: Acuvue Advance — Silicone hydrogel contact lens

SUMMARY:
The purpose of this study is to compare the performance of the ACUVUE® ADVANCE® Plus lenses against ACUVUE® ADVANCE® lenses in the plus power parameters.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be at least 18 years of age and no more than 45 years of age.
* The subject is a current spherical soft contact lens wearer and willing to wear the study lenses on a daily wear basis for the duration of the study (defined as a minimum of 6 hours with a minimum of at least 1 month's wear prior to the study).
* The subject's optimal verified spherical equivalent distance correction must be between +1.00 and + 6.00D.
* Any cylinder power must be ≤ 0.75D.
* The subject must have visual acuity best correctable to 20/25+3 or better for each eye.
* The subject must read and sign the Statement of Informed Consent.
* The subject must appear able and willing to adhere to the instructions set forth in the clinical protocol.

Exclusion Criteria:

* Ocular or systemic allergies or disease which might interfere with contact lens wear.
* Systemic disease or use of medication which might interfere with contact lens wear.
* Clinically significant (grade 3 or 4) corneal edema, corneal vascularization, corneal staining, or any other abnormalities of the cornea which would contraindicate contact lens wear.
* Clinically significant (grade 3 or 4) tarsal abnormalities or bulbar injection which might interfere with contact lens wear.
* Any ocular infection.
* Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
* Pregnancy or lactation.
* Diabetes.
* Infectious diseases (e.g. hepatitis, tuberculosis) or an immuno-suppressive disease (e.g. HIV).
* Habitual contact lens type is toric, bifocal, in monovision contact lens wear, or is worn as extended wear.
* Need any near correction.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Winter Park, Florida
  - New York, New York
  - Nanticoke, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a 3 site, 3 visit, randomized, double-masked, bilateral crossover trial comparing Acuvue Advance to Acuvue Advance Plus lenses.
Pre-assignment Details: Of the 38 subjects enrolled, 2 were ineligible and not-randomized, 3 discontinued, and 33 completed as cohort.
Groups:
- Acuvue Advance Plus/ Acuvue Advance; Acuvue Advance/ Acuvue Advance Plus: Group 1 wore AAP first and AA second. Group 2 wore AA first and AAP second
Period: Baseline
Arm/Group | Acuvue Advance Plus/ Acuvue Advance | Acuvue Advance/ Acuvue Advance Plus
Started | 18 | 18
Completed | 17 | 16
Not Completed | 1 | 2
Not completed — Lack of Efficacy | 1 | 2
Period: 1-Week Follow-Up
Arm/Group | Acuvue Advance Plus/ Acuvue Advance | Acuvue Advance/ Acuvue Advance Plus
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0
Period: Final Visit
Arm/Group | Acuvue Advance Plus/ Acuvue Advance | Acuvue Advance/ Acuvue Advance Plus
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline summary was conducted on subjects who successfully completed the study. There were 38 subjects that started, 3 discontinued, and 2 were ineligible.
Groups:
- All Subjects: Subjects who were randomized and successfully completed the study.
Arm/Group | All Subjects
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (5.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Visual Acuity One Week After Lens Wear
Description: Visual acuity was measured using ETDRS visual acuity test. ETDRS stands for Early Treatment Diabetic Retinopathy Study. Binocular and monocular measurements were collected.
Time Frame: 1 week
Population: Subjects analyzed were those who were enrolled, randomized, and completed the study. Both monocular and binocular measurements were taken and included in analysis.
Measure: Least Squares Mean (Standard Error); unit: LogMAR
Units Other Than Participants: eyes
Groups:
- Acuvue Advance Plus: Acuvue Advance Plus contact lenses-Binocular measurements
- Acuvue Advance: Acuvue Advance contact lenses - Binocular Measurements
Arm/Group | Acuvue Advance Plus | Acuvue Advance
Number analyzed (Participants) | 33 | 33
Number analyzed (eyes) | 66 | 66
LogMAR
  Low Luminance/ High Contrast (Binocular) | 0.11 (0.082) | 0.10 (0.063)
  Low Luminance/ High Contrast (Monocular) | 0.14 (0.100) | 0.14 (0.088)
  High Luminance/ Low Contrast (Binocular) | 0.12 (0.075) | 0.13 (0.067)
  High Luminance/ Low Contrast (Monocular) | 0.22 (0.108) | 0.21 (0.097)
Statistical Analysis 1: Comparison: Acuvue Advance Plus vs Acuvue Advance; For Low Luminance/ High Contrast grouping (Monocular): Ho: The test lens (Acuvue Advance Plus) will be non-inferior to the control lens (Acuvue Advance). Ha: The test lens (Acuvue Advance Plus) will be <= to the control lens (Acuvue Advance); Test type: Non-Inferiority or Equivalence — Non-inferiority is assessed with a margin of -0.05logMAR; Mixed Models Analysis; Mean Difference (Final Values) = 0.007, 95% CI 2-sided [-0.0044 to 0.0187], Standard Error of Mean 0.0059 — The mean difference is defined by: Test lens (Acuvue Advance Plus) - control lens (Acuvue Advance)
Statistical Analysis 2: Comparison: Acuvue Advance Plus vs Acuvue Advance; High Luminance/ Low Contrast grouping (Binocular): Ho: The test lens (Acuvue Advance Plus) will be non-inferior to the control lens (Acuvue Advance). Ha: The test lens (Acuvue Advance Plus) will be <= to the control lens (Acuvue Advance); Test type: Non-Inferiority or Equivalence — Non-inferiority is assessed with a margin of -0.05 logMAR; Mixed Models Analysis; Mean Difference (Final Values) = 0.003, 95% CI 2-sided [-0.0086 to 0.0146], Standard Error of Mean 0.0059 — The mean difference is defined by: Test lens (Acuvue Advance Plus) - control lens (Acuvue Advance)

2. Primary Outcome: Visual Acuity at Time of Initial Fit
Description: Visual acuity will be measured using ETDRS visual acuity test. ETDRS stands for Early Treatment Diabetic Retinopathy Study.
Time Frame: After 10-15 minutes of lens wear
Population: Analysis is conducted on those were enrolled and completed the trial.
Measure: Mean (Standard Deviation); unit: LogMAR
Units Other Than Participants: eyes
Groups:
- Acuvue Advance Plus: Acuvue Advance Plus contact lenses worn
- Acuvue Advance: Acuvue Advance contact lenses worn
Arm/Group | Acuvue Advance Plus | Acuvue Advance
Number analyzed (Participants) | 33 | 33
Number analyzed (eyes) | 66 | 66
LogMAR
  Low Luminance/High Contrast (Binocular) | 0.13 (0.087) | 0.11 (0.073)
  Low Luminance/High Contrast (Monocular) | 0.16 (0.106) | 0.15 (0.101)
  High Luminance/Low Contrast (Binocular) | 0.14 (0.076) | 0.13 (0.094)
  High Luminance/Low Contrast (Monocular) | 0.24 (0.123) | 0.21 (0.111)
Statistical Analysis 1: Comparison: Acuvue Advance Plus vs Acuvue Advance; For Low Luminance/ High Contrast Grouping (Monocular): Ho: The test lens (Advance Plus) will be non-inferior to the control lens (Advance). Ha: The test lens (Advance Plus) will be <= to the control lens (Advance); Test type: Non-Inferiority or Equivalence — Non-inferiority is assessed with a margin of -0.05 logMAR; Mixed Models Analysis; Mean Difference (Final Values) = 0.016, 95% CI 2-sided [0.0041 to 0.0282], Standard Error of Mean 0.0061 — Mean difference represents: Test lens (Advance Plus) - Control lens (Advance)
Statistical Analysis 2: Comparison: Acuvue Advance Plus vs Acuvue Advance; For High Luminance/ Low Contrast Grouping (Binocular): Ho: The test lens (Advance Plus) will be non-inferior from the control lens (Advance). Ha: The test lens (Advance Plus) will be <= to the control lens (Advance); Test type: Non-Inferiority or Equivalence — Non-inferiority is assessed with a margin of -0.05 logMAR; Mixed Models Analysis; Mean Difference (Final Values) = 0.021, 95% CI 2-sided [0.0090 to 0.3305], Standard Error of Mean 0.006 — Mean Difference is defined to be: test lens (Advance Plus) - control lens (Advance)

3. Secondary Outcome: Contact Lens Comfort Using Contact Lens User Experience (CLUE)
Description: The subjective comfort questionnaire CLUE, assesses the overall lens comfort. The CLUE Questionnaire is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0 to 120.
Time Frame: 1 week
Population: Analysis was on those who were enrolled and completed the study.
Measure: Least Squares Mean (Standard Error); unit: CLUE points
Arm/Group | Acuvue Advance Plus | Acuvue Advance
Number analyzed (Participants) | 33 | 33
CLUE points | 49.2 (3.28) | 50.7 (3.26)

4. Secondary Outcome: Subject Reported Vision Using Contact Lens User Experience (CLUE).
Description: Overall vision was assessed by a subjective vision questionnaire. The CLUE Questionnaire is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0 to 120.
Time Frame: 1 week
Population: Analysis was on those who were enrolled and completed the study.
Measure: Least Squares Mean (Standard Error); unit: CLUE points
Arm/Group | Acuvue Advance Plus | Acuvue Advance
Number analyzed (Participants) | 33 | 33
CLUE points | 42.5 (2.87) | 39.9 (2.86)

5. Secondary Outcome: Contact Lens Comfort at Initial Fit Using Contact Lens User Experience (CLUE)
Description: Comfort was assessed using a subjective comfort questionnaire. The CLUE Questionnaire is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. CLUE scores have a range of 0-120.
Time Frame: Baseline
Population: Analysis was on those who were enrolled and completed the study.
Measure: Least Squares Mean (Standard Error); unit: CLUE points
Arm/Group | Acuvue Advance Plus | Acuvue Advance
Number analyzed (Participants) | 33 | 33
CLUE points | 65.3 (3.14) | 59.0 (3.19)

6. Secondary Outcome: Subject Reported Vision at Initial Fit Using Contact Lens User Experience (CLUE)
Description: Vision at initial fit was assessed using a subjective vision questionnaire. The CLUE Questionnaire is a validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0 to 120.
Time Frame: Baseline
Population: Subjects analyzed included only those who were enrolled and completed the study.
Measure: Least Squares Mean (Standard Error); unit: CLUE points
Arm/Group | Acuvue Advance Plus | Acuvue Advance
Number analyzed (Participants) | 33 | 33
CLUE points | 46.7 (3.90) | 49.6 (3.98)

ADVERSE EVENTS:
Time Frame: 1 month, Study took place from Oct 1, 2010-Nov 12, 2010
Groups:
- Acuvue Advance Plus: Acuvue Advance Plus contact lenses
- Acuvue Advance: Acuvue Advance contact lenses
Arm/Group | Acuvue Advance Plus | Acuvue Advance
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days